CLINICAL TRIAL: NCT01715727
Title: Diagnosis of Parkinson's Disease Using Diffusion Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Wang . Jiun-Jie (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Wang . Jiun-Jie, Associate Professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: 100-3761A3
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson Disease
Keywords: diffusion kurtosis imaging; parkinson disease; parkinsonism; diagnosis; differential diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Parkinson's Disease for follow-up: 1. Patients should fulfill the National Institute of Neurological Disorders and Stroke in USA ( NINDS ) Diagnostic Criteria for Parkinson Disease(37) for "probable" PD, except for the age of onset.
  2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
  3. Able to understand and provide signed informed consent.
  4. Early to moderate stage defined as Hohen and Yahr stage 1-3,
- Parkinsons"s Disease with severity match: Parkinsons"s Disease with severity match: 30 subjects
  1. Patients should fulfill the National Institute of Neurological Disorders and Stroke in USA ( NINDS ) Diagnostic Criteria for Parkinson Disease(37) for "probable" PD, except for the age of onset.
  2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
  3. Able to understand and provide signed informed consent.
  4. Severity matched with PSP (subjects = 15)/MSA (subjects= 15), the severity was judged by Hohen and Yahr stage
- Healthy age matched controls: Healthy age matched controls: subjects = 112
  1. Healthy subjects without a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.
  2. Able to understand and provide signed informed consent.
  3. Age range and gender matched with Parkinsons"s Disease for follow up.
- Parkinson Plus Syndrome Group M: 1. MSA Patients should fulfill the NINDS Consensus statement for the clinical diagnosis of probable MSA
  2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
  3. Able to understand and provide signed informed consent
- Parkinson Plus Syndrome Group P: 1. PSP Patients should fulfill the NINDS-SPSP and Litvan criteria(4) for probable PSP
  2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
  3. Able to understand and provide signed informed consent.

SUMMARY:
The hypothesis of the study is that the dopaminergic cell death located in the basal ganglia of the brain in patients with Parkinson's Disease can be detected by diffusion Magnetic Resonance Imaging, specifically by diffusion kurtosis imaging. The preliminary result was published in Radiology 2011. The current study proposed to investigate the following issues:

* validation of diagnostic sensitivity and specificity
* differential diagnosis capability between PD and PD+ syndrome
* prognosis capability

In the first year, patients with Parkinson's disease will be recruited from the outpatient clinics of movement disorders in ChangGung memorial hospital Linkou, Taiwan. The diffusion parameters in basal ganglia will be compared with a group of healthy controls. In the second year, patients with progressive supranuclear palsy and patients with multiple system atrophy will be recruited for assessment of differential diagnosis. The patients with Parkinson's Disease will return for assessment of disease severity and in the third year, for the outcome evaluation.

DETAILED DESCRIPTION:
Currently there existed no specific diagnostic test of Parkinson's Disease. Accurate diagnosis is of great interest because of the reduction in health cost and disease co-morbidity, improvement in effective treatment course and avoidance of un-necessary intervention. Our preliminary result showed superior performance from diffusion kurtosis imaging, a new development in MRI since 2007, on the diagnosis of Parkinson's Disease when compared to conventional diffusion MRI. The study proposes to validate the diagnostic value of diffusion kurtosis in major basal ganglia regions using a cross-sectional study and to assess the prognostic value through 3-year longitudinal follow-up. Furthermore, the iron content as well as global white matter involvement in both PD and PD plus syndrome patients will be assessed. The difference in MRI information between PD and PD plus syndrome patients will then be addressed in a comprehensive manner.

One hundred and twelve patients with Parkinson's Disease will be recruited in the first year and followed up for 3 years. Another 112 healthy controls will be included. This is to validate the diagnosis and assess the prognosis. Another 30 patients with Parkinson's Disease, 15 patients with progressive supranuclear palsy and 15 patients with multiple system atrophy will be recruited in the 2nd year for differential diagnosis. The imaging protocol will include both diffusion tensor and diffusion kurtosis imaging. Susceptibility weighted imaging will be included for iron content estimation. The targeted anatomy will include regional changes in basal ganglia, midbrain as well as thalamus, and global white matter changes using tract based spatial statistics. The statistical analysis will use receiver operative characteristics to assess the diagnostic performance, Spearman's ranked correlation for correlation with disease severity and net reclassification improvement for differential diagnosis. The prognostic value will be determined by the decline rate and the quality of life.

The end points of the project are to differentiate patients of PD from PD plus syndrome, and to predict the clinical outcomes using diffusion MRI. Patent application will be filed in the first year. The analysis of medical device software and software life cycle processes and the evaluation of risk management to medical devices will be filed at the end of the third year.

ELIGIBILITY:
Inclusion Criteria:

Parkinsons"s Disease for follow up: 112 subjects

1. Patients should fulfill the National Institute of Neurological Disorders and Stroke in USA ( NINDS ) Diagnostic Criteria for Parkinson Disease(37) for "probable" PD, except for the age of onset.
2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
3. Able to understand and provide signed informed consent. 4. Early to moderate stage defined as Hohen and Yahr stage 1-3, subjects = 100

Parkinsons"s Disease with severity match: 30 subjects

1. Patients should fulfill the National Institute of Neurological Disorders and Stroke in USA ( NINDS ) Diagnostic Criteria for Parkinson Disease(37) for "probable" PD, except for the age of onset.
2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
3. Able to understand and provide signed informed consent. 4. Severity matched with PSP (subjects = 15)/MSA (subjects= 15), the severity was judged by Hohen and Yahr stage

Healthy age matched controls: subjects = 112 1. Healthy subjects without a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness. 2. Able to understand and provide signed informed consent. 3. Age range and gender matched with Parkinsons"s Disease for follow up.

Parkinson Plus Syndrome Group M ( Multi System Atrophy, subjects = 15 ):

1. MSA Patients should fulfill the NINDS Consensus statement for the clinical diagnosis of probable MSA(38) 2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours. 3. Able to understand and provide signed informed consent 2012/04/20 第二版 14

Parkinson Plus Syndrome Group P (Progressive Supranuclear Palsy, subjects = 15):

1. PSP Patients should fulfill the NINDS-SPSP and Litvan criteria(4) for probable PSP
2. Able to tolerate the disability during the "drug-off" state, at least for 12 hours.
3. Able to understand and provide signed informed consent.

Exclusion Criteria:

The following exclusion criteria apply to all groups.

1. Cardiac pacemaker implantation.
2. Implantation of intracranial metal device.
3. Significant major systemic disease, such as renal failure, heart failure, stroke, AMI/unstable angina, poor controlled diabetes mellitus, poor controlled hypertension.
4. Pregnant or breast feeding women.
5. Moderate to severer dementia.
6. Severe dyskinesia
7. Any documented abnormality of brain in the brain by MRI and 18FDG PET studies, which might contribute to the cognitive function, such as hydrocephalus or encephalomalacia, will be excluded. Mild cortical atrophy will be allowed.
8. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
9. Significant physical disorder or neuropsychiatric disorder.
10. Except the medication for parkinsonism and related symptoms, subjects who received any medication that can pass the blood-brain barrier will be excluded.
11. Except the medication for parkinsonism and related symptoms, subjects who chronically take any drug for more than 10 years will be excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the movement disorder clinics in ChangGung memorial hospital LinKou. The healthy control will be recruited from the local community in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
differential diagnosis | end of the second year
  To differentiate patient of PD from PD + using diffusion MRI

SECONDARY OUTCOMES:
prognosis | end of the third year
  To predict the outcome of patient with PD using the diffusion MRI at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jiun-Jie Wang, PhD, Principal Investigator — ChangGung University
Locations (1):
- ChangGung Memorial Hospital, Linkou, Taoyuan, Taiwan, Taiwan

REFERENCES:
- [Background] Wang JJ, Lin WY, Lu CS, Weng YH, Ng SH, Wang CH, Liu HL, Hsieh RH, Wan YL, Wai YY. Parkinson disease: diagnostic utility of diffusion kurtosis imaging. Radiology. 2011 Oct;261(1):210-7. doi: 10.1148/radiol.11102277. Epub 2011 Jul 19. PMID 21771952